CLINICAL TRIAL: NCT06385496
Title: MATCH Treatment Subprotocol L: Phase II Study of MLN0128 (TAK-228) in Patients With Tumors Wtih mTOR Mutations
Brief Title: Testing MLN0128 (TAK-228) as Potentially Targeted Treatment in Cancers With mTOR Genetic Changes (MATCH - Subprotocol L)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2024-01145; NCI-2024-01145 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); EAY131-L; EAY131-L (Other: ECOG-ACRIN Cancer Research Group); EAY131-L (Other: CTEP); U10CA180820 (NIH)
Record Dates: First submitted 2024-04-25; First posted 2024-04-26 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Advanced Lymphoma; Advanced Malignant Solid Neoplasm; Refractory Lymphoma; Refractory Malignant Solid Neoplasm; Refractory Multiple Myeloma
MeSH Terms: conditions — Lymphoma; Multiple Myeloma | interventions — Biopsy; Specimen Handling; Magnetic Resonance Spectroscopy; sapanisertib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (sapanisertib [MLN0128 (TAK-228)]) (Experimental): Patients receive sapanisertib (MLN0128 [TAK-228]) PO QD on days 1-28 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo CT or MRI during screening and on study, as well as during follow-up as clinically necessary. Patients also undergo biopsies and blood sample collection on study.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Drug: Sapanisertib

INTERVENTIONS:
Procedure: Biopsy Procedure — Undergo biopsy
  Other Names: Biopsy; BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Drug: Sapanisertib — Given PO
  Other Names: INK-128; INK128; MLN-0128; MLN0128; TAK-228

SUMMARY:
This phase II MATCH treatment trial tests how well MLN0128 (TAK-228) works in treating patients with cancer that has certain genetic changes called mTOR mutations. MLN0128 (TAK-228) may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the proportion of patients with objective response (OR) to targeted study agent(s) in patients with advanced refractory cancers/lymphomas/multiple myeloma.

SECONDARY OBJECTIVES:

I. To evaluate the proportion of patients alive and progression free at 6 months of treatment with targeted study agent in patients with advanced refractory cancers/lymphomas/multiple myeloma.

II. To evaluate time until death or disease progression. III. To identify potential predictive biomarkers beyond the genomic alteration by which treatment is assigned or resistance mechanisms using additional genomic, ribonucleic acid (RNA), protein and imaging-based assessment platforms.

IV. To assess whether radiomic phenotypes obtained from pre-treatment imaging and changes from pre- through post-therapy imaging can predict objective response and progression free survival and to evaluate the association between pre-treatment radiomic phenotypes and targeted gene mutation patterns of tumor biopsy specimens.

OUTLINE:

Patients receive sapanisertib (MLN0128 [TAK-228]) orally (PO) once daily (QD) on days 1-28 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo computed tomography (CT) or magnetic resonance imaging (MRI) during screening and on study, as well as during follow-up as clinically necessary. Patients also undergo biopsies and blood sample collection on study.

After completion of study treatment, patients are followed every 3 months for 2 years and then every 6 months for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have met applicable eligibility criteria in the Master MATCH Protocol EAY131/ NCI-2015-00054 prior to registration to treatment subprotocol
* Patients must fulfill all eligibility criteria of MATCH Master Protocol at the time of registration to treatment step (Step 1, 3, 5, 7)
* Patients must have a mutation in mTOR, KEAP1 or NFE2L2 as determined via the MATCH Master Protocol
* Patients must have an electrocardiogram (ECG) within 8 weeks prior to treatment assignment and must NOT have any of the following cardiac criteria:

  * Clinically important abnormalities in rhythm, conduction or morphology of resting ECG (e.g. complete left bundle branch block, third degree heart block, Corrected QT Interval [QTc] interval > 480 milliseconds)
  * Uncontrolled hypertension (i.e., systolic blood pressure >180 mm Hg, diastolic blood pressure > 95 mm Hg). Use of anti-hypertensive agents to control hypertension before cycle 1, day 1 is allowed
  * Known pulmonary hypertension.
* Patients must not have known hypersensitivity to MLN0128 or compounds of similar chemical or biologic composition
* Patients must not have known hepatitis B surface antigen-positive, or known or suspected active hepatitis C infection, but may have had previously treated and successfully eradicated hepatitis C virus (HCV)
* Patients must have none of the following within six months of receiving the first dose of MLN0128 (TAK-228): ischemic, myocardial or cerebrovascular event, class III or IV heart failure, placement of pacemaker, or pulmonary embolism
* Patients must have no manifestations of malabsorption due to prior gastrointestinal (GI) surgery, GI disease, or for an unknown reason that may alter the absorption of MLN0128 (TAK-228)
* Patients who have a history of brain metastasis are eligible for the study provided that all the following criteria are met:

  * Brain metastases which have been treated
  * No evidence of disease progression for >= 1 months before the first dose of study drug
  * No hemorrhage after treatment
  * Off-treatment with dexamethasone for 4 weeks before administration of the first dose of MLN0128 (TAK-228)
* No ongoing requirement for dexamethasone or anti-epileptic drugs
* Patients meeting the following criteria for concomitant medications prior to starting MLN0128 (TAK-228) are not eligible for the study:

  * Patients who use a proton pump inhibitor (PPI) within 7 days before receiving the first dose of study drug.
  * Patients who would require treatment with PPIs throughout the trial
  * Patients who would need to take H2 receptor antagonists within 24 hours of the first dose of study drug NOTE Strong CYP1A2 inhibitors and CYP inducers should be administered with caution, at the discretion of the investigator. Alternative treatments, if available, should be considered
* Patients must not have known treatment with systemic corticosteroid within one week prior to the first administration of study drug
* Patients must not have uncontrolled diabetes mellitus. Controlled diabetes is defined as: Glycosylated hemoglobin (HbA1c) < 7.0%, or fasting serum glucose (=< 130 mg/dL)
* Patients must not have fasting triglycerides >= 300 mg/dL
* Patients must not have had prior treatment with other known TORC1/2 inhibitors, including:

  * AZD8055
  * XL765
  * BEZ235
  * GSK2126458
  * XL388
  * DS3078(a)
  * PF-05212384
  * SF1126
  * Palomid-529
  * GDC0980 (apitolisib)
  * LY30223414
  * BKM120
  * OSI0127
  * MLN0128 (TAK-228)
  * AZD2014
* Patients must not have other clinically significant co-morbidities that, in the opinion of the investigator, would limit compliance with study requirements
* Fertility and developmental studies with MLN0128 (TAK-228) have not been conducted. On the basis of potential hazard of other mTOR inhibitors (i.e., rapamycin and other rapalogs) on the developing fetus, women of childbearing age should avoid becoming pregnant while taking MLN0128 (TAK-228). For this reason, women of child-bearing potential and men must agree to practice 1 highly effective method of contraception and 1 additional effective (barrier) method of contraception, at the same time, from the time of signing the informed consent through 120 days after the last dose of study drug, or agree to completely abstain from heterosexual intercourse. Men must agree not to donate sperm during the course of this study or within 120 days after receiving their last dose of study drug
* Patients who are known to be HIV-positive are not eligible for this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2017-03-12 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Up to 3 years
  ORR is defined as the percentage of patients whose tumors have a complete or partial response to treatment among analyzable patients. Objective response is defined consistent with Response Evaluation Criteria in Solid Tumors version 1.1, the Cheson (2014) criteria for lymphoma patients, and the Response Assessment in Neuro-Oncology criteria for glioblastoma patients. 90% two-sided confidence interval is calculated for ORR. For the purposes of this study, patients should be re-evaluated for response:
  * For treatments given in 21 day (3 week) cycles: every 3 cycles (9 weeks) for the first 33 cycles, and every 4 cycles thereafter (12 weeks)
  * For treatments given in 28 day (4 week) cycles: every 2 cycles (8 weeks) for the first 26 cycles, and every three cycles thereafter (12 weeks)
  * For treatments given in 42 day (6 week) cycles: every 2 cycles (12 weeks)

SECONDARY OUTCOMES:
Overall survival (OS) | From start of treatment on that step until death, or censored at the date of last contact, assessed up to 3 years
  Will be evaluated specifically for each drug (or step). OS will be estimated using the Kaplan-Meier method.
6-month progression free survival (PFS) | From start of treatment on that step until determination of disease progression or death from any cause, censored at the date of last disease assessment for patients who have not progressed, assessed at 6 months
  Progression free survival is defined as time from treatment start date to date of progression or death from any cause, whichever occurs first. Disease progression was evaluated using the Response Evaluation Criteria in Solid Tumors version 1.1, the Cheson (2014) criteria for lymphoma patients, and the Response Assessment in Neuro-Oncology criteria for glioblastoma patients. Please refer to the protocol for detailed definitions of disease progression. 6 month PFS rate was estimated using the Kaplan-Meier method, which can provide a point estimate for any specific time point.
Progression free survival | From start of treatment on that step until determination of disease progression or death from any cause, censored at the date of last disease assessment for patients who have not progressed, assessed up to 3 years
  PFS was defined as time from treatment start date to date of disease progression or death from any causes, whichever occurred first. Median PFS was estimated using the Kaplan-Meier method. Disease progression was evaluated using the Response Evaluation Criteria in Solid Tumors version 1.1, the Cheson (2014) criteria for lymphoma patients, and the Response Assessment in Neuro-Oncology criteria for glioblastoma patients. Please refer to the protocol for detailed definitions of disease progression.

CONTACTS AND LOCATIONS:
Overall Officials: John L Hays, Principal Investigator — ECOG-ACRIN Cancer Research Group
Locations (1):
- ECOG-ACRIN Cancer Research Group, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.]
URL: https://grants.nih.gov/policy/sharing.htm